CLINICAL TRIAL: NCT00823147
Title: Pain Catastrophizing as a Cause for Systemic Inflammation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Darnall, PhD (Other)
Collaborators: Oregon Clinical and Translational Research Institute (Other); Office of Research on Women's Health (ORWH) (NIH)
Responsible Party: Sponsor-Investigator, Beth Darnall, PhD, Principal Investigator, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 4920; 5 K12 HD04348807
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Musculoskeletal Pain
Keywords: Pain; Systemic Inflammation; Pain Catastrophizing
MeSH Terms: conditions — Musculoskeletal Pain; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pain Catastrophizing Induction Group (Experimental): Collect salivary cortisol kit if subject did not mail from home Full battery of self-report measures given. Pain ratings taken (0-10). Height and weight measured. Heart monitor affixed. Catheter placed; 25 minute rest.
  Catastrophizing group: 10-minute catastrophizing induction. Participants self-rate their level of emotional distress.
  Subsequent blood draws occur per protocol time points:
  1. 25 minutes following IV placement (BASELINE)
  2. 15 minutes post catastrophizing induction (stress experiment)
  3. 90 minutes (1.5 hours) post-induction
  4. 150 minutes (2.5 hours) post-induction
  5. 210 minutes (3.5 hours) post-induction
  6. 270 minutes (4.5 hours) post-induction
  Interventions: Behavioral: Pain Catastrophizing Induction
- Control Group (No Intervention): Collect salivary cortisol kit if subject did not mail from home Full battery of self-report measures given. Pain ratings taken (0-10). Height and weight measured. Heart monitor affixed. Catheter placed; 25 minute rest.
  Control group: Persons in this group will rest, complete puzzles, read emotionally-neutral material or watch videos provided to them.
  Blood draws and saliva samples gathered per protocol time points:
  1. 25 minutes following IV placement (BASELINE- T1)
  2. 25 minutes following baseline T2
  3. 115 minutes (1 hour 55 min) post baseline T3
  4. 175 minutes (2 hours 55 min) post baseline T4
  5. 235 minutes (3 hours 55 min) post baseline T5
  6. 295 minutes (4 hours 55 min) post baseline T6

INTERVENTIONS:
Behavioral: Pain Catastrophizing Induction — Participants will undergo a psychologist-guided 10-minute induction of negative cognitive focus on the theoretical future worsening of one's pain condition.Biological stress response will be measured via heart rate, blood pressure and serum cortisol.
  Arms: Pain Catastrophizing Induction Group

SUMMARY:
Research shows that the immune system is involved in chronic pain. The immune system is involved in the process of inflammation. The investigators are still learning about the factors that cause inflammation, but know it can be measured in the blood. The purpose of this study is to understand how negative thoughts affect the immune system in women with chronic pain.

A sub-study asks subjects to store a blood sample for future research by the PI aimed at identifying genetic markers in women with chronic pain.

DETAILED DESCRIPTION:
A main goal of the study is to better understand pain mechanics. Research has linked pro-inflammatory cytokines to the development and progression of pain. Research has also linked female gender with increases in pro-inflammatory cytokines (relative to males) following psychological stress. Therefore, we hypothesize that women in the study who evidence significantly increased pro-inflammatory cytokines following pain catastrophizing may be at risk for the progression of their pain condition.

The sample will be 60 women having chronic musculoskeletal pain (we will enroll up to 75 persons to account for attrition and screen failures but require the usable data of only 60 women). Based on enrollment rates for our previous study, and given our expanded catchment area, we expect to enroll 60 persons within approximately 14 months and to complete the experimental phase of the study within approximately 17 months. The follow-up phase of the study will continue, for as long as participants agree to be followed for up to 10 years.

The study design is a randomized, controlled experiment. Participants are consented and enrolled under the impression that they will undergo one stress experiment day (lasting about 5.5 hours). However, on their study day we will randomize subjects to either be in the control group or the catastrophizing (stress) group.

Screening Visit: The purpose of this visit is to determine eligibility and obtain informed consent. Inclusion and exclusion criteria will be assessed through medical record review, a screening interview, and a hormonal bloodspot kit. A questionnaire will also be given to determine level of depressive symptoms and to assess for suicidality. The hormonal bloodspot kit involves a finger prick and obtaining about 5-6 drops of blood. If lab analysis of this kit determines abnormal hormonal levels, persons will be excluded from further participation in the study. Participants will be given a saliva kit to gather 4 saliva samples at home over the course of one day. Participants will store these saliva samples in their refrigerator. They will either bring in the kit at the time of their study visit or mail the kit in a prepaid box given to them (the hormones in the saliva are shelf stable for up to 3 weeks; we will ask participants to refrigerate the samples if they are not immediately mailing them or bringing them to the study site. In this way we will best ensure that samples will be preserved and usable). All participants enrolled in the study will be under the impression that they will be participating in a catastrophizing experiment during their study day. However, only half of the participants will actually experience the 10-minute stress experiment on experiment day. We have included this minor form of deceit in the protocol so we can control for the anticipatory stress of expecting to experience a negative emotional experiment. We highlight here that the mild deception will occur for only half the sample (those going into the control group) and it represents a decrease in risk for these persons.

Study Visit: This study visit is scheduled to occur during the follicular phase of the menstrual cycle (this phase follows the menstrual period and is easy to predict in our sample of normally menstruating women by using a calendar). If difficulty is encountered in predicting the date of the follicular phase, participants will call the PI or study coordinator when their menstrual period begins to schedule their study date (approximately 5-6 days from onset on menses). All participants arrive in a fasting state, during their follicular phase to control for sex-steroid influences on immunity. 3ml of blood will be drawn for hormone levels. The hormone level will not be analyzed at this time, but saved until the end of the study for analysis, if needed. A complete cardiometabolic panel will be measured via bloodspot. If the subject agrees to take part in the sub study, we will take an additional 10mL of blood for an extra bloodspot card that we will store for future pain/genomic research. Pain ratings will be assessed, and questionnaires will be completed. Standardized meals (with no caffeine) will be served to participants (breakfast, lunch, snacks). An OCTRI research nurse will place an intravenous catheter into the arm of participant's choosing. A Holter heart monitor will be placed on participants by nursing. This is a portable device that measures heart beat. Placement of the leads around the heart involves cleaning the skin. The monitor will remain affixed for the duration of the study visit. At this point participants will be randomized to either be in the control group or in the catastrophizing group using a random number generator. After they are randomized into one of the two groups, the deception will be revealed to the control group, and its rationale explained. Those randomized to the stress group will be informed of the deception, and the rationale for having used it, at the conclusion of the study visit .

Those in the control group will have serum measurements taken at the time points listed in the study activities table below. They will occupy themselves for the next 4.5 hours with activity options to keep them from sleeping during the study visit, such as reading magazines, crossword puzzles, or games. We will have these on hand, or they can bring them to the visit. At each time point, salivary cortisol, heart rate, blood pressure, and pain ratings will be assessed. At the end of the final blood draw, the IV catheter is removed and the first study visit is complete.

Those persons randomized to the catastrophizing group will undergo a 10min pain catastrophizing induction following the 25 min post- IV catheterization rest period (we are also calling this the stress experiment). The PI will guide participants to focus on their pain, to imagine it worsening in the near future, and to describe how their worsening pain will affect life domains most important to them. The induction is standardized in the following ways: 1) duration of induction (10 minutes); 2) imaginal focus on pain worsening in the near future; 3) participants are guided to describe the anticipated negative consequences of their pain worsening; 4) participants will be guided to describe the ways in which they feel helpless while imagining the scenario. Items 2-4 are designed to tap the 3 components of pain catastrophizing (rumination, magnification of pain, helplessness).

Pain ratings and stress response will be measured via heart rate and blood pressure and salivary cortisol according to the study activities table below. No bloodspot kits will be collected during this visit. This study visit ends after the 270min post-induction blood draw. The PI will debrief subjects and assess their affective state. Free counseling will be offered before the subject leaves the study visit (only one person in the previous study opted for the post-study counseling). If anyone in the stress group would like a counseling referral the PI will provide local options to them. All participants receive a next-day telephone call to assess for mood state and adverse events.

Long-term Follow-Up: We have included a separate consent form to allow us to follow subjects over time. A main goal of the study is to better understand pain mechanics. Research has linked pro-inflammatory cytokines to the development and progression of pain. Research has also linked female gender with increases in pro-inflammatory cytokines (relative to males) following psychological stress. Therefore, we hypothesize that women in the study who evidence significantly increased pro-inflammatory cytokines following pain catastrophizing may be at risk for the progression of their pain condition. We expect that if we follow our sample over time, we will see a trend that will serve as preliminary data to allow us to investigate this further. While the catastrophizing experiment will provide us with meaningful data, this longitudinal sub study will allow us to define the clinical and functional relevance of our findings. For those who consent to this related study, subjects will be contacted every 6 months for up to 10 years and asked several questions about their pain, mood, function, and stress levels. They will also be asked to complete 4 questionnaires including: the Oswestry Disability Index, The CES-D form, and the Perceived Stress Scale. These questionnaires can be read to the subject over the phone or completed on paper. If the subject would like to complete them on paper, an address, stamped return envelope will be provided. They will also be asked if we can contact them again in 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages 18-70
* Non-smokers
* Diagnosed with musculoskeletal chronic pain
* Normal menstrual cycle or postmenopausal

Exclusion Criteria:

* Psychosis or suicidality
* Current Major Depression
* Former intravenous drug user
* Needle/blood/injection phobia
* Limited venous access
* Sex-steroid dysregulation
* Self-Reported Pregnancy
* Fibromyalgia or inflammatory disease, e.g. lupus
* Active corticosteroid regimen
* Taking beta blockers
* Taking oral contraception or hormone therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2009-01; Primary Completion 2012-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in pro-inflammatory cytokine levels assessed from immunoassay samples | 3.5 hours
Change in anti-inflammatory cytokine levels assessed from immunoassay samples | 3.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Beth Darnall, Ph.D, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science Universtiy, Portland, Oregon, United States